CLINICAL TRIAL: NCT07375030
Title: Evaluation of Patient-specific Surgical Stents and Plates for Guided Reduction And Fixation of Mandibular Angle Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00010824-12/2023
Record Dates: First submitted 2026-01-17; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Mandibular Angle Fracture
Keywords: Mandibular angle fracture; guided reduction and fixation
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with recent mandibular angle fractures managed with patient specific stents and plates (Experimental)
  Interventions: Device: Patient specific surgical stents and plates for guided reduction and fixation of mandibular angle fixation

INTERVENTIONS:
Device: Patient specific surgical stents and plates for guided reduction and fixation of mandibular angle fixation — Patient specific surgical stents and plates for guided reduction and fixation of mandibular angle fixation

SUMMARY:
This study will evaluate the patient specific surgical stent and plate for guided reduction and fixation of mandibular angle fractures.

DETAILED DESCRIPTION:
seven patients with recent mandibular angle fractures indicated for open reduction and internal fixation were treated by patient specific surgical stent and plate for guided reduction and fixation of mandibular angle fractures. Follow-up extended to 12 weeks. Clinical parameters included pain, operative time, postoperative occlusion, wound healing and mouth opening. Radiographic evaluation was conducted using computed tomography scans acquired preoperatively and postoperatively ,superimposition of the pre and postoperative models will be done to create error map and measure the accuracy

ELIGIBILITY:
Inclusion Criteria:

* Medically fit patients free from relevant conditions contraindicating surgery.
* Patients with mandibular angle fracture indicated for open reduction and internal fixation.
* Presented within 2 weeks from trauma.

Exclusion Criteria:

* Infected fracture site.
* Patients with systemic bone diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of accuracy of surgical reduction and fixation | Day 1
  Evaluation of accuracy of surgical guide will be done using slicer and blender, and mimics software with the aid of the preoperative and postoperative CT. Preoperative planning will be merged with the new CT data to identify the accuracy of reduction.

SECONDARY OUTCOMES:
Clinical evaluation for Intra-opreative time | Intra-opreative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes